CLINICAL TRIAL: NCT07393828
Title: Efficacy of Biofilm Removal of Different Interproximal Oral Hygiene Devices Around Posterior Single Implants in Peri-Implant Mucositis: A Randomized Clinical Trial
Brief Title: Effectiveness of Interproximal Cleaning Devices for Biofilm Removal Around Posterior Single Implants With Peri-Implant Mucositis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PER-ECL-2025-04
Record Dates: First submitted 2026-01-21; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Peri-implant Mucositis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interdental Brush Group (Experimental): Participants use interdental brushes for interproximal plaque control around posterior implants.
  Interventions: Device: Participants assigned to this intervention group are instructed to perform daily interproximal plaque control around implant-supported crowns using the allocated interdental oral hygiene device (inter
- Oral Irrigator Group (Experimental): Participants use an oral irrigator for interproximal plaque control around posterior implants.
  Interventions: Device: Participants assigned to this intervention group are instructed to perform daily interproximal plaque control around implant-supported crowns using the allocated interdental oral hygiene device (inter
- Superfloss Group (Experimental): Participants use Superfloss for interproximal plaque control around posterior implants.
  Interventions: Device: Participants assigned to this intervention group are instructed to perform daily interproximal plaque control around implant-supported crowns using the allocated interdental oral hygiene device (inter

INTERVENTIONS:
Device: Participants assigned to this intervention group are instructed to perform daily interproximal plaque control around implant-supported crowns using the allocated interdental oral hygiene device (inter — Participants will receive a structured oral hygiene intervention using interproximal oral hygiene devices specifically designed for use around posterior single implants diagnosed with peri-implant mucositis. The intervention consists of standardized instruction and supervised use of the assigned interproximal device according to manufacturer recommendations and a predefined clinical protocol. The device will be used by participants for daily interproximal plaque control around the implant site throughout the study period. Clinical and microbiological outcomes related to biofilm accumulation and peri-implant soft tissue inflammation will be assessed at predefined follow-up visits. No pharmacological agents are administered as part of the intervention.

SUMMARY:
This randomized clinical trial aims to evaluate and compare the efficacy of different interproximal oral hygiene devices for biofilm removal around posterior single dental implants in patients diagnosed with peri-implant mucositis.

Peri-implant mucositis is a reversible inflammatory condition of the peri-implant soft tissues caused primarily by bacterial biofilm accumulation. Effective plaque control is essential for the prevention of disease progression to peri-implantitis. However, there is limited clinical evidence regarding the comparative effectiveness of different interproximal oral hygiene devices in implant-supported sites.

A total of approximately 75 patients with posterior single implants and peri-implant mucositis will be recruited. Participants will be randomly allocated to one of the study groups, each using a specific interproximal oral hygiene device as part of their daily oral hygiene regimen. All participants will receive standardized oral hygiene instructions at baseline.

Clinical parameters related to peri-implant inflammation and plaque accumulation will be assessed at baseline and at follow-up visits at 1, 3, and 6 months. The primary outcome is the reduction of peri-implant biofilm accumulation. Secondary outcomes include changes in clinical inflammatory parameters around the implants.

The results of this study are expected to provide clinically relevant evidence to support evidence-based recommendations for interproximal oral hygiene in patients with dental implants affected by peri-implant mucositis.

ELIGIBILITY:
Inclusion Criteria:

Adults aged ≥18 years. Presence of at least one posterior single dental implant in function for ≥12 months.

Diagnosis of peri-implant mucositis, defined as bleeding on probing with probing depths ≤5 mm and no radiographic bone loss beyond initial remodeling.

Good general health (ASA I-II). Ability and willingness to comply with study procedures and follow-up visits. Provision of written informed consent.

Exclusion Criteria:

Diagnosis of peri-implantitis (radiographic bone loss beyond initial remodeling).

Uncontrolled systemic diseases affecting periodontal or peri-implant health (e.g., uncontrolled diabetes mellitus).

Use of systemic antibiotics or anti-inflammatory drugs within the previous 3 months.

Current pregnancy or lactation. Current smoker of >10 cigarettes/day. History of periodontal therapy or professional implant maintenance within the previous 3 months.

Use of medications known to affect bone metabolism (e.g., bisphosphonates). Inability to perform adequate oral hygiene or to attend scheduled study visits.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in peri-implant biofilm accumulation | Baseline (pre-intervention) to 1month post-intervention, 3 months post-intervetion, 6 months post-intervention
  Change in interproximal peri-implant biofilm accumulation measured using a validated plaque index (e.g., Modified Plaque Index) at posterior single implants.
Change in peri-implant biofilm accumulation | Baseline (pre-intervention) to 1month post-intervention, 3 months post-intervetion, 6 months post-intervention
  The primary outcome measure is the change in peri-implant biofilm accumulation following the use of the assigned interproximal oral hygiene device. Biofilm levels will be assessed at implant-supported posterior sites using a validated plaque index specific for peri-implant tissues. Measurements will be recorded at baseline and after the intervention period, and the difference between time points will be used for analysis.

SECONDARY OUTCOMES:
Change in peri-implant probing pocket depth | Baseline (pre-intervention) to 1month post-intervention, 3 months post-intervetion, 6 months post-intervention
  This secondary outcome assesses changes in peri-implant probing pocket depth (PPD) following the use of different interproximal oral hygiene devices. Probing depth will be measured at standardized peri-implant sites using a calibrated periodontal probe, and changes from baseline will be analyzed to evaluate the clinical response of peri-implant tissues.